CLINICAL TRIAL: NCT02770625
Title: A Multicenter, Open-Label Phase III Study to Evaluate the Safety and Efficacy of ISU302 (Imiglucerase for Injection) in Patients With Type 1 Gaucher Disease
Brief Title: Phase III Study of ISU302 in Patients With Type 1 Gaucher Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ISU Abxis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISU302-004
Record Dates: First submitted 2016-05-07; First posted 2016-05-12 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-02

CONDITIONS: Gaucher Disease, Type 1
Keywords: Type I Gaucher; ISU302; Imiglucerase
MeSH Terms: conditions — Gaucher Disease | interventions — imiglucerase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ISU302 (Experimental): 60 U/kg (once every 2 weeks for 6 months)
  Interventions: Drug: ISU302

INTERVENTIONS:
Drug: ISU302 — 60 U/kg given intravenously
  Other Names: Imiglucerase

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ISU302 in patients with Type 1 Gaucher disease.

DETAILED DESCRIPTION:
The objectives of this clinical study were to evaluate the efficacy and safety of every other week (EOW) dosing of ISU302 at a dose of 60 U/kg as an effective glucocerebrosidase enzyme replacement therapeutic product in patients with Type 1 Gaucher disease (GD). Primary efficacy endpoint was the difference in hemoglobin concentration between baseline and Week 24. Secondary efficacy endpoints included assessment of platelet counts, spleen and liver volume, and biomarker levels in plasma at Week 24 compared to baseline; skeletal change and bone mineral density (BMD); and single-dose pharmacokinetic (PK) analysis. Secondary safety endpoints included the assessment of adverse events (AEs), vital signs, physical examination, and electrocardiogram (ECG); clinical safety laboratory analyses included serum chemistry, urinalysis, hematology and coagulation, and the measurement of anti-ISU302 antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 GD.
* Documented glucocerebrosidase deficiency.
* GD-related anemia, defined as hemoglobin levels of at least 1 g/dL below the lower limit of normal for age and gender and one or more of the following 3 criteria:

  * At least moderate splenomegaly (2 to 3 cm below the left costal margin) by palpation,
  * GD-related thrombocytopenia, defined as a platelet count <90 x 109 platelets/L,
  * GD-related readily palpable enlarged liver.
* Not received treatment for GD (investigational products, miglustat, velaglucerase alfa, or imiglucerase) within 12 months prior to study entry.
* Ability to comprehend and willing to sign the ICF.
* Legal guardian (and patient if age appropriate) understood the nature of the procedure, was willing to comply with associated follow-up evaluations, and provided written informed consent and assent prior to the procedure.
* Female patients of childbearing potential must had agreed to use a medically acceptable method of contraception at all the times during the study. Male patients must have used a medically acceptable method of birth control throughout their participation in the study and were required to report the pregnancy of a partner.

Exclusion Criteria:

* Type 2 or 3 GD.
* Splenectomy.
* Antibody positive to ISU302 or imiglucerase during screening or the patient had experienced an anaphylactic reaction to ISU302 or imiglucerase. - Treatment with any non-GD-related investigational drug or medical device within 30 days prior to study entry; such use during the study was also not permitted.
* Currently receiving red blood cell (RBC) growth factor (eg, erythropoietin) chronic systemic corticosteroids or received such treatment within the last 6 months.
* Positive for human immunodeficiency virus (HIV) and hepatitis B or C.
* Exacerbated anemia at screening (due to iron, folic acid, or vitamin B12 deficiency or infectious/immune-mediated cause).
* Significant comorbidity(ies) that could affect study data or confounded the study results (eg, malignancies, primary biliary cirrhosis, autoimmune liver disease).
* Pregnant or lactating female patients and those not willing to use highly effective barrier or medical method of contraception.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amel El Beshlawy, Prof., Principal Investigator — Abou El Reesh Children's Hospital

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 9 patients were planned to be enrolled in the study; 8 patients were enrolled into the study and all 8 patients completed the study.
Period: Overall Study
Arm/Group | ISU302
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ISU302
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.8 (4.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 8
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)] | 17.244 (1.9236)
Weight [Mean (Standard Deviation); unit: kg] | 17.9 (7.64)
Height [Mean (Standard Deviation); unit: cm] | 100.40 (22.852)

OUTCOME MEASURES:

1. Primary Outcome: The Difference in Hemoglobin Concentration [g/dL]
Time Frame: from baseline to Week 24
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | ISU302
Number analyzed (Participants) | 7
g/dL
  Baseline | 9.49 (0.857)
  Visit 13 (Week 24) | 11.44 (0.870)

2. Secondary Outcome: Platelet Counts [10^3 Platelets/uL]
Time Frame: from baseline to Week 24
Measure: Mean (Standard Deviation); unit: 10^3 platelets/uL
Arm/Group | ISU302
Number analyzed (Participants) | 7
10^3 platelets/uL
  Baseline | 132.6 (72.27)
  Visit 13 (Week 24) | 180.3 (47.10)

3. Secondary Outcome: Spleen Volume
Time Frame: from baseline to Week 24
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | ISU302
Number analyzed (Participants) | 7
Milliliters
  Baseline | 29.047 (18.9140)
  Visit 13 (Week 24) | 15.207 (9.4730)

4. Secondary Outcome: Liver Volume
Time Frame: from baseline to Week 24
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | ISU302
Number analyzed (Participants) | 7
Milliliters
  Baseline | 1.530 (0.6078)
  Week 24 | 1.537 (0.5059)

5. Secondary Outcome: Angiotensin-converting Enzyme Level
Time Frame: from baseline to Week 24
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ISU302
Number analyzed (Participants) | 7
U/L
  Baseline | 195.71 (108.952)
  Week 24 | 159.31 (58.253)

6. Secondary Outcome: Chitotriosidase Level (Nmol/mL/hr)
Time Frame: from baseline to Week 24
Measure: Mean (Standard Deviation); unit: nmol/mL/hr
Arm/Group | ISU302
Number analyzed (Participants) | 7
nmol/mL/hr
  Baseline | 11093.67 (10354.369)
  Visit 13 (Week 24) | 3409.63 (3103.006)

7. Secondary Outcome: Chemokine Ligand (CCL-18) Level [ng/mL]
Time Frame: from baseline to Week 24
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ISU302
Number analyzed (Participants) | 7
ng/mL
  Baseline | 927.05 (595.4552)
  Week 24 | 577.331 (310.0457)

8. Secondary Outcome: Acid Phosphatase (ACP) Level (U/L)
Time Frame: from baseline to Week 24
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ISU302
Number analyzed (Participants) | 7
U/L
  Baseline | 25.44 (7.517)
  Week 24 | 15.44 (4.313)

9. Secondary Outcome: Skeletal Status Improvement
Description: The number of participant who have the skeletal status diagnosed as Osteosclerosis
Time Frame: from baseline to Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | ISU302
Number analyzed (Participants) | 7
Participants
  Baseline | 7
  Week 24 | 7

10. Secondary Outcome: Change in Bone Mineral Density
Time Frame: from baseline to Week 24
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | ISU302
Number analyzed (Participants) | 7
g/cm^2
  Baseline | -0.954 (1.5967)
  Week 24 | -0.104 (2.4558)

11. Other Pre Specified Outcome: Assessment of AEs, Vital Signs, Physical Examination, and Electrocardiogram (ECG)
Time Frame: Screening to Visit14 (Week 26)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years and 4 months
Arm/Group | ISU302
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISU302 (N=8)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Bronchitis / Infections and infestations
Viral pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pneumonia viral / Infections and infestations
Ludwig angina (Cardiac disorders) | 1 (1) — Ludwig angina / Infections and infestations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes